CLINICAL TRIAL: NCT01358214
Title: Single-center, Non-randomized, Comparative, Post-marketing Surveillance Cohort Study on Validation of a Questionnaire on Quality of Life After Surgical Stabilization of the Urethra With Titanized Polypropylene Mesh (TiLOOP® Tape)
Brief Title: Quality of Life After Tension Free Transvaginal Sling / Tape Operation With a Titanized Surgical Tape (TiLOOP® Tape)
Status: Terminated | Type: Observational
Why Stopped: major recruitment failure
Sponsor: pfm medical gmbh (Industry)
Collaborators: Aix Scientifics (Industry)
Responsible Party: Sponsor
Other Study IDs: pfm 10k003 TiLOOP® Tape
Record Dates: First submitted 2011-05-18; First posted 2011-05-23 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Urinary Incontinence, Stress
Keywords: Sub-urethral Sling; Treatment Outcome; Quality of Life
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients treated with a surgical mesh: This arm of study patients is defined by patients treated with a TiLOOP® Tape mesh between 2007 and 2009 at the Franziskus Krankenhaus, Berlin. The sample of the treated population represents the patient population for which the medical device is intended. To minimize selection bias without compromising patients' rights and welfare, all treated patients will be invited. These patients will be asked to participate in the validation of the questionnaire on quality of life. In addition to this safety and effectiveness of the surgical mesh implantation will be collected
  Interventions: Behavioral: Questionnaire on Quality of Life.
- Intended to be treated with a mesh: This arm of the study populations is defined by patients in whom a clinical anamnesis independent of the requirements of this study suggests that a sub-urethral sling operation is indicated. These patients will be asked to participate in the validation of the questionnaire on quality of life.
  Interventions: Behavioral: Questionnaire on Quality of Life.
- Non-symptomatic Population: This arm of the study population is defined by women that show no symptoms of incontinence. They will be asked to participate in the validation of the questionnaire on quality of life.
  Interventions: Behavioral: Questionnaire on Quality of Life.

INTERVENTIONS:
Behavioral: Questionnaire on Quality of Life. — The impact of a disease on patient's Quality of Life has meanwhile gained more influences on the choice of treatment alternatives. The benefit of a method is currently not only defined by the objective outcome but also influenced by the Quality of Life. Two questionnaires with 20 respectively 40 Questions should be filled in by the patients.
  Other Names: QoL

SUMMARY:
Validation of a new Quality of Life (QoL) questionnaire in a population of patient gaining a TiLOOP® TAPE surgical mesh for stabilization of the urethra.

DETAILED DESCRIPTION:
The prevalence of urinary incontinence in the adult female population has been estimated between 10% and 40%. Several treatment alternatives have been suggested until now. Nevertheless, the ideal treatment has not been identified yet. On the one hand this is related to the low amount of valid scientific information regarding different treatment methods. On the other hand the impact of patients' quality of life, which plays a major role, has not been fully considered. To date, there is no established Questionnaire on Quality of Life that provides physicians an assistance to obtain information on the subjective effects caused by stress urinary incontinence.

In the present study the patients' Quality of Life will be assessed by use of two questionnaires, that is a new one and an already validated questionnaire. The study population consists of patients who already received an implantation of a sub-urethral surgical mesh (TiLOOP® Tape), of symptomatic patients before an operation, and of a group of non-symptomatic women. Subjects will be asked in a single visit only to fill in both questionnaires.

Furthermore the safety and effectiveness of the TiLOOP® Tape mesh will be evaluated in the study arm of treated patients.

Study has been terminated after major recruitment failure (only 21 instead of 240 patients has been included).

ELIGIBILITY:
Inclusion Criteria:

* Depending on study arm:
* Women with a TiLOOP® Tape implant, Implanted between 2007 and 2009 at the study center - OR -
* Woman with a planned Tape implantation at the study center - OR -
* Woman with no disease related to incontinence
* Subject is able to understand the nature, relevance and significance of the clinical trial
* Subject has given informed consent

Exclusion Criteria:

* Subject revoked consent
* Lack of subject's compliance regarding data collection or examination in the scope of the trial (Non-Compliance)
* Subject institutionalized by court or official order (MPG §20.3)
* Subject participates in another clinical investigation

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The indicated or treated population of women showing stress urinary incontinence that should / has been treated with a surgical mesh.
  The sample of patients treated with TiLOOP® Tape at the single center between 2007 and 2009 represents the patient population for which the medical device is intended. The clinic continues to examine women with incontinence symptoms requiring a mesh implant. This group of patients is assumed to be similar to the study arm of treated patients.
  The Non-symptomatic Population consists of women comparable in age but without urinary incontinence
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2011-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Validation of a new questionnaire on quality of life | before treatment (baseline) or 6 to 24 months after treatment, respectively
  It is expected that the newly developed questionnaire on quality of life (QoL) is equal or better in description of the impact on QoL regarding the differentiation of the study populations, as compared to the standard questionnaire.

SECONDARY OUTCOMES:
Safety of surgical mesh implantation for treatment of urinary incontinence | 6-24 months after treatment
  In the study arm of treated patients the study outcome will describe all safety relevant events occurred within the period from implantation until scheduled study examination. The time between scheduled examination and implantation varies as the implantation it not part of this study. The findings will therefore be stratified by 6 months, 12 months and 24 months after implantation.
Effectiveness of surgical mesh implantation for treatment of urinary incontinence | 6-24 months after treatment
  In the study arm of treated patients, the study outcome will describe the efficacy of the TiLOOP® Tape implantation based on successful implantation and complications observed during the period from implantation until discharge from the hospital. The time between scheduled examination and implantation varies as the implantation it not part of this study. The findings will therefore be stratified by 6 months, 12 months and 24 months after implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Beer, Prof. MD, Principal Investigator — Franziskus-Krankenhaus Berlin Akademisches Lehrkrankenhaus der Charité - Universtätsmedizin Berlin
Locations (1):
- Franziskus-Krankenhaus Berlin Akademisches Lehrkrankenhaus der Charité - Universtätsmedizin Berlin, Berlin, Germany